CLINICAL TRIAL: NCT05131490
Title: Effect on Physical and Psychosocial Adaptation of Mobile Application Developed for Gynecological Cancer Patients Receiving Chemotherapy
Brief Title: Effect on Adaptation to Cancer of Mobile Application Developed for Gynecological Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Okan Vardar, Lecturer, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 60116787-020/34123
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Gynecologic Cancer; Chemotherapy Effect; Mobile Application; Physiological Adaptation; Psychosocial Adaptation
Keywords: Gynecologic Cancer; Chemotherapy Effect; Mobile Application; Physiological Adaptation; Psychosocial Adaptation

STUDY DESIGN:
Intervention Model Description: Single blind pre-post test randomized controlled design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental group intervention consists two months a mobile application intervention developed for gynecological cancer patients receiving chemotherapy
  Interventions: Behavioral: A mobile application intervention developed for gynecological cancer patients receiving chemotherapy
- No intervention (No Intervention): Control group receive routine care.

INTERVENTIONS:
Behavioral: A mobile application intervention developed for gynecological cancer patients receiving chemotherapy — The mobile application will consist of modules. It is planned to include four education modules and consultancy modules in the application.
  1. Module 1: It will consist of sub-categories with information to be prepared in line with the current literature on gynecological cancer types and treatments applied. There will be information and short videos that will strengthen coping with physical symptoms, especially from chemotherapy.
  2. Module 2: In this area, there will be meditation and relaxation/breathing exercises, information on relaxing complementary therapies, anxiety reduction and stress management techniques videos and audio recordings.
  3. Module 3: Current developments on gynecological cancers will be included.
  4. Module 4: Encouraging recovery stories and videos of cancer survivors will be included.
  5. Module 5: Counseling module. This is the area where patients who cannot find answers in the frequently asked questions section can ask questions to the research team.
  Arms: Experimental

SUMMARY:
Getting a cancer diagnosis, the difficult treatments applied and the side effects that occur completely affect the life of the patient, shaking his future plans and adaptation mechanisms. In recent years, the role of healthcare professionals has included counseling and promoting positive health behaviors to reduce disease and treatment side effects and increase adherence to disease. The service provided by healthcare professionals to patients has started to move to digital environments with the developing technology and the concept of e-health has been born. Offering e-health support as part of regular care has become a powerful tool to help cancer patients manage their disease. Web-based interventions or mobile applications provide an opportunity for improved communication and better information exchange between healthcare professionals and patients. In addition, education of cancer patients and patient self-management allow for better clinical outcomes using e-health or mobile health applications. The widespread use of smartphones enables cancer patients to be supported from different perspectives through mobile applications. When the studies are examined, it is noteworthy that mobile applications developed for female cancer patients are predominantly related to breast cancer. Most of the technology-based researches on gynecological cancers are studies conducted through text message intervention, online web-based interventions or social media tools such as Facebook and WeChat. For this reason, the aim of this study is to develop a mobile application to increase physical and psychosocial adjustment for gynecological cancer patients receiving chemotherapy and to investigate its effectiveness.

DETAILED DESCRIPTION:
This study was planned as a parallel, single-blind, pre-post-test randomized controlled experimental study in which two groups (experiment-control) will be compared. The block randomization method will be used. The patients who will participate in the research will be reached through social media networks related to cancer (Facebook and Instagram account of the Dance with Cancer Association, etc.) and the data will be collected from patients who are suitable for the sample characteristics through mobile application. The sample size was calculated in the G*power statistics program by utilizing the data of a study in which on cancer patients using a mobile application intervention was previously performed (α =0.05, d=0.75). Accordingly, it was found that 23 people should be taken for each group to sampling for 80% power. Considering that there might be losses, the number of samples was increased by 10% and it was planned to include a total of 52 people in the study. Intention-to-treat analysis will be performed to manage bias and losses.

A pilot application will be conducted for 4 weeks with 6 patients regarding the usability of the mobile application and these patients will not be included in the study. At the end of 4 weeks, feedback will be received from the patients participating in the pilot application with the mobile application evaluation form. Necessary changes will be made in the mobile application in line with the feedback.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Be at least primary school graduate
* Volunteering to participate in research
* Being diagnosed with gynecological cancer for the first time (no cancer recurrence)
* Receiving at least one course of chemotherapy and continuing chemotherapy treatment
* Be Eastern Cooperative Oncology Group (ECOG) performance scale score below 3
* Be not have a psychiatric illness
* Owning a smartphone
* Be have internet access and have used any mobile application before

Exclusion Criteria:

* Be have any psychiatric illness
* Be have not yet received or completed chemotherapy treatment
* Be Eastern Cooperative Oncology Group (ECOG) performance scale score of 3 and above

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with gynecological cancer
Enrollment: 64 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
The Psychosocial Adjustment to İllnes Scale-Self Report (PAIS-SR) | Change from baseline PAIS-SR score at 4 and 8 weeks
  The scale measures the interaction of individuals with other individuals and institutions forming the socio-cultural environment and consists of 7 sub-dimensions. These; Health Care Orientation (8 items); Vocational Environment (6 items); Domestic Environment (8 items); Sexual Relationship (6 items); extended family relationships (5 items); social environment (6 items); psychological pressure (7 items) it consists of 46 items in total, including. It is calculated by giving scores ranging from 0 to 3 for the items in the scale. Major negative changes since illness are scored with 3 points, no change or positive changes with 0 points. A score below 35 indicates "good psychosocial adjustment", a score between 35 and 51 indicates "moderately good psychosocial adjustment", and a score above 51 indicates "poor psychosocial adjustment". An increase in the score is an indication of difficulty in adaptation and deterioration.
MD Anderson Symptom Inventory (MDASI) | Change from baseline MDASI score at 4 and 8 weeks
  It is a short inventory that measures the impact and severity of cancer-related symptoms. Each symptom is evaluated at 11 levels (0=no symptoms, 10=very bad).
  The scale consists of two sub-dimensions and 19 items. In the first part of the inventory, "symptoms" (13 items), in the second part "inhibition of the individual's life" (6 items) and the situation in the last 24 hours are evaluated. In the event that the life of the individual in the second part of the inventory is hindered; general activity, mood, work and/or works in home, relationships with other people, walking, enjoying life are evaluated. A high score indicates an increase in the severity of the symptom and a negative impact on life.
Hospital Anxiety and Depression Scale (HADS) | Change from baseline HADS score at 4 and 8 weeks
  The aim of the scale is not to diagnose, but to determine the risk group by scanning anxiety and depression in a short time in patients with physical illness. The scale has anxiety (HADS-A) and depression (HADS-D) subscales. The scale is a self-report scale and consists of 14 items, 7 of which investigate symptoms of anxiety and 7 of which investigate symptoms of depression. Responses are evaluated on a four-point Likert scale and scored between 0-3. Odd numbers measure anxiety, even numbers measure depression.
  For both subscales, "7 and below" non-patients, "8-10" borderline patients, and "11 and above" patient evaluations were deemed appropriate. The scoring of each item in the scale is different. Items 1, 3, 5, 6, 8, 10, 11, and 13 show decreasing severity and the scoring is 3, 2, 1, 0. On the other hand, the 2nd, 4th, 7th, 9th, 12th and 14th items are scored as 0, 1, 2, 3, respectively. The lowest score that can be obtained from both subscales is 0, and the highest score is 21.
Assessment of Survivor Concerns (ASC) | Change from baseline ASC score at 4 and 8 weeks
  The scale was developed in 2007 to evaluate the fear of recurrence of cancer and general health in cancer patients. The scale has two subscales: "cancer worry subscale" and "general health worry subscale". The scale included six items and three in each subscale. However, as the sixth item was 'children's health worry"' which cannot be administered to those who have no children, the scale was revised, and this item was removed. The number of items was reduced to five. The new 5-item form of the scale is recommended. According to the revised scale, the "cancer worry subscale" is comprised of three items and the "general health scale" two items. The Assessment of Survivor Concerns Scale is a 4-point Likert type scale that is evaluated as "not at all" and "very much". The lowest score possible on this scale is five and the highest is 20. Higher scores indicate higher levels of concern.
Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline
  The ECOG Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). This numbering scale is one way to define the population of patients to be studied in the trial. The scale was developed by the Eastern Cooperative Oncology Group (ECOG), now part of the ECOG-ACRIN Cancer Research Group, and published in 1982. It is used to promote greater standardization among researchers who design and evaluate clinical cancer studies and to assess the general well-being of patients. A score between 0 and 5 is made.
Mobile Application Evaluation Form | At the end of the 4-week pilot application
  It is a form created by researchers to evaluate satisfaction with the use of the mobile application. With this form, after the "pilot application" from patients will receive feedback on the ease of use and content of the mobile application.
Introductory Information Form | Baseline
  It is the form that contains information about the socio-demographic characteristics of the patients diagnosed with gynecological cancer and the type, duration and stage of the diagnosed gynecological cancer, the treatments received and the number of chemotherapy cycles.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)